CLINICAL TRIAL: NCT03577262
Title: A Non-therapeutic Feasibility Study to Evaluate the Kinetics and Test-retest Repeatability and Reproducibility of the Radioligand [11C]-UCB-J for Imaging Synaptic Density in Healthy Subjects and Mild-to-moderate Alzheimer's Disease Subjects
Brief Title: A Non-therapeutic Feasibility Study of the Radioligand [11C]-UCB-J for Imaging Synaptic Density
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Collaborators: QPS Netherlands B.V. (Industry); University Medical Center Groningen (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RDN-NI-001
Record Dates: First submitted 2018-05-24; First posted 2018-07-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one

STUDY DESIGN:
Intervention Model Description: evaluate the kinetics and test-retest repeatability and reproducibility of the radioligand [11C]-UCB-J for imaging synaptic density in up to10 healthy subjects and then mild to moderate Alzheimer's Disease patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects [11C]-UCB-J (Experimental): Net dose of approximately 370 megabecquerel (MBq) of [11C]-UCB-J, Total injected mass of UCB-J per will not to exceed 10 µg for each dose given on Days 1 and 28
  Interventions: Other: [11C]-UCB-J
- AD patients [11C]-UCB-J (Experimental): Net dose of approximately 370 megabecquerel (MBq) of [11C]-UCB-J, Total injected mass of UCB-J per will not to exceed 10 µg for each dose given on Days 1 and 28
  Interventions: Other: [11C]-UCB-J

INTERVENTIONS:
Other: [11C]-UCB-J — IV radioligand given prior to and during positron emission tomography (PET) scan

SUMMARY:
Up to 20 subjects will receive an injection with [11C]-UCB-J followed by a PET scan on Days 1 and 28

DETAILED DESCRIPTION:
After assessing eligibility during a 4-week screening period, approximately 20 subjects will participate in the PET acquisition phase of the study. Drop-outs or unevaluable subjects will be replaced for a target sample size of 20 completed and evaluable subjects.

During the screening period, a 3D T1-weighted MRI must be acquired and reviewed for exclusion criteria and acquisition quality.

On the day of radioligand administration (Day 1), subjects will come to the study center for an ambulatory visit (Visit 1). After re-confirming eligibility, all subjects will receive an injection with [11C]-UCB-J followed by a PET scan.

Using an arterial line and manual sampling, blood samples will be collected up to 90 minutes after radioligand injection in order to quantify radioactivity concentration in whole blood and plasma as well as parent fraction over time.

Subjects will return to the clinic for one more ambulatory visit on Day 28 ± 3 (Visit 2). The same procedures will be performed as on Day 1.

PET scanning duration will be initially set to 90 minutes. After a minimum of 4 subjects have completed baseline and Day 28 scans, 90 minute and 60 minute scan data will be analyzed. Based on this analysis, and at the discretion of the investigator, it will be decided whether the remaining subjects will require 60 or 90 minute scans.

Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Healthy male or female age 55 - 75 years old, inclusive, at the time of informed consent.
* Mini-mental state examination (MMSE) greater than or equal to 27.

Group 2

* Adult males or females age 55 - 75 years old, inclusive, at the time of informed consent.
* Confirmed diagnosis of mild-to-moderate AD, defined as:

  1. National Institute on Aging - Alzheimer's Association (NIA-AA) "probable" diagnosis (see Appendix 2);
  2. MMSE 18-26.

Exclusion Criteria:

* History or current evidence of any clinically significant cardiovascular, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic (with the exception of AD in Group 2), psychiatric, renal, or other major disease, as determined by the Investigator.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Measure [11C]-UCB-J plasma radioactivity levels in plasma over time | Day 1 to 28
Measure concentration of radioactivity as a function of time according to pre-defined brain regions | Day 1 to 28

CONTACTS AND LOCATIONS:
Overall Officials: Coordinating PI, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - VU Medical Center, Dept. Radiology and Nuclear Medicine, Amsterdam
  - QPS Netherlands B.V., Groningen
  - University Medical Center Groningen, Nuclear Medicine and Molecular Imaging, Groningen

IPD SHARING:
Plan to Share IPD: No